CLINICAL TRIAL: NCT00005504
Title: Longitudinal Investigation of Thromboembolism Etiology
Brief Title: Epidemiology of Venous Thrombosis and Pulmonary Embolism
Acronym: LITE
Status: Active, not recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 9701M12240; R01HL059367 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Cardiovascular Diseases; Pulmonary Embolism; Venous Thrombosis
MeSH Terms: conditions — Cardiovascular Diseases; Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, serum, plasma
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
To investigate venous thromboembolism in two carefully conducted prospective epidemiologic studies of African American and white adults -- the Atherosclerosis Risk in Communities (ARIC) Study and the Cardiovascular Health Study (CHS).

DETAILED DESCRIPTION:
BACKGROUND:

Venous thromboembolism, comprising deep venous thrombosis (DVT) and pulmonary embolism (PE), is a major contributor to morbidity and mortality in the United States. Nevertheless, no comprehensive, prospective, population-based epidemiologic studies have simultaneously examined lifestyle, molecular, and biochemical risk factors for this important disease.

DESIGN NARRATIVE:

Deep venous thrombosis and pulmonary embolism cases were identified and verified in order to estimate incident rates of hospitalized venous thromboembolism in the combined ARIC and CHS cohorts. The association of venous thromboembolism was determined prospectively with demographic and lifestyle factors, plasma lipids, medical history, and hemostatic components (including fibrinogen, platelet count, factors VIIc and VIIIc) using existing ARIC and CHS data. A nested case control study was conducted using stored pre-diagnosis blood and DNA specimens to determine the prospective associations of venous thromboembolism with the following: levels of procoagulant or anticoagulant factors and related genetic variants (including factor V Leiden), fibrinolytic factors (e.g., plasminogen activator inhibitor-1) and related genetic variants, markers of thrombin activation, and other potentially important biochemical or related genetic factors (e.g., homocysteine).

The study was renewed in 2003 to extend event follow-up for four more years and to conduct longitudinal analyses of incidence and potential risk factors not fully explored such as diet, frailty, hormone replace therapy and obesity interactions. It was renewed in 2008 to conduct a genome wide association study. It was again renewed in 2013 and 2017.

ELIGIBILITY:
Inclusion: in the ARIC or CHS cohorts already

Exclusion: not in the ARIC or CHS cohorts

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ARIC and CHS cohorts
Sampling Method: Probability Sample
Enrollment: 21680 (Actual)
Dates: Start 1998-02 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Venous thrombosis and pulmonary embolism | Yearly Follow up
  venous thrombosis and pulmonary embolism

CONTACTS AND LOCATIONS:
Overall Officials: Weihong Tang, PhD, Principal Investigator — University of Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Folsom AR, Aleksic N, Wang L, Cushman M, Wu KK, White RH. Protein C, antithrombin, and venous thromboembolism incidence: a prospective population-based study. Arterioscler Thromb Vasc Biol. 2002 Jun 1;22(6):1018-22. doi: 10.1161/01.atv.0000017470.08363.ab. PMID 12067914
- [Background] Folsom AR, Cushman M, Tsai MY, Aleksic N, Heckbert SR, Boland LL, Tsai AW, Yanez ND, Rosamond WD. A prospective study of venous thromboembolism in relation to factor V Leiden and related factors. Blood. 2002 Apr 15;99(8):2720-5. doi: 10.1182/blood.v99.8.2720. PMID 11929758
- [Background] Folsom AR, Cushman M, Tsai MY, Heckbert SR, Aleksic N. Prospective study of the G20210A polymorphism in the prothrombin gene, plasma prothrombin concentration, and incidence of venous thromboembolism. Am J Hematol. 2002 Dec;71(4):285-90. doi: 10.1002/ajh.10229. PMID 12447958
- [Background] Folsom AR, Cushman M, Heckbert SR, Rosamond WD, Aleksic N. Prospective study of fibrinolytic markers and venous thromboembolism. J Clin Epidemiol. 2003 Jun;56(6):598-603. doi: 10.1016/s0895-4356(03)00052-0. PMID 12873656
- [Background] Aleksic N, Folsom AR, Cushman M, Heckbert SR, Tsai MY, Wu KK. Prospective study of the A455V polymorphism in the thrombomodulin gene, plasma thrombomodulin, and incidence of venous thromboembolism: the LITE Study. J Thromb Haemost. 2003 Jan;1(1):88-94. doi: 10.1046/j.1538-7836.2003.00029.x. PMID 12871544
- [Background] Tsai AW, Cushman M, Tsai MY, Heckbert SR, Rosamond WD, Aleksic N, Yanez ND, Psaty BM, Folsom AR. Serum homocysteine, thermolabile variant of methylene tetrahydrofolate reductase (MTHFR), and venous thromboembolism: Longitudinal Investigation of Thromboembolism Etiology (LITE). Am J Hematol. 2003 Mar;72(3):192-200. doi: 10.1002/ajh.10287. PMID 12605391
- [Background] Tsai AW, Cushman M, Rosamond WD, Heckbert SR, Tracy RP, Aleksic N, Folsom AR. Coagulation factors, inflammation markers, and venous thromboembolism: the longitudinal investigation of thromboembolism etiology (LITE). Am J Med. 2002 Dec 1;113(8):636-42. doi: 10.1016/s0002-9343(02)01345-1. PMID 12505113
- [Background] Cushman M, Tsai AW, White RH, Heckbert SR, Rosamond WD, Enright P, Folsom AR. Deep vein thrombosis and pulmonary embolism in two cohorts: the longitudinal investigation of thromboembolism etiology. Am J Med. 2004 Jul 1;117(1):19-25. doi: 10.1016/j.amjmed.2004.01.018. PMID 15210384
- [Background] Fashanu OE, Heckbert SR, Aguilar D, Jensen PN, Ballantyne CM, Basu S, Hoogeveen RC, deFilippi C, Cushman M, Folsom AR. Galectin-3 and Venous Thromboembolism Incidence: the Atherosclerosis Risk in Communities (ARIC) Study. Res Pract Thromb Haemost. 2017 Oct;1(2):223-230. doi: 10.1002/rth2.12038. Epub 2017 Sep 4. PMID 29152608
- [Background] Folsom AR, Tang W, George KM, Heckbert SR, MacLehose RF, Cushman M, Pankow JS. Prospective study of gamma' fibrinogen and incident venous thromboembolism: The Longitudinal Investigation of Thromboembolism Etiology (LITE). Thromb Res. 2016 Mar;139:44-9. doi: 10.1016/j.thromres.2016.01.008. Epub 2016 Jan 12. PMID 26916295
- [Background] Folsom AR, Tang W, Weng LC, Roetker NS, Cushman M, Basu S, Pankow JS. Replication of a genetic risk score for venous thromboembolism in whites but not in African Americans. J Thromb Haemost. 2016 Jan;14(1):83-8. doi: 10.1111/jth.13193. Epub 2015 Dec 29. PMID 26565658